CLINICAL TRIAL: NCT02785224
Title: Arterial Pressure and Stress-Dose Steroids in In-hospital Cardiac Arrest: a Mediation Analysis of Prior Randomized Clinical Trial Data.
Brief Title: Arterial Pressure and Stress-Dose Steroids in Cardiac Arrest.
Status: Withdrawn | Type: Observational
Why Stopped: No funding could be obtained for this study
Sponsor: University of Athens (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, MD, PhD, DEAA, EDIC, Associate Professor of Intensive Care Medicine, University of Athens
Other Study IDs: AP-MEDIATION-15516/23/5/16
Record Dates: First submitted 2016-05-22; First posted 2016-05-27 (Estimated); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vasopressin Steroids Epinephrine (VSE): Patients with in-hospital cardiac arrest treated with vasopressin, methylprednisolone, and epinephrine during cardiopulmonary resuscitation, and also with stress-dose hydrocortisone for postresuscitation shock.
  Interventions: Drug: Vasopressin Steroids Epinephrine
- Control: Patients with in-hospital cardiac arrest treated with normal saline placebo, normal saline placebo, and epinephrine during cardiopulmonary resuscitation, and also with normal saline placebo for postresuscitation shock.

INTERVENTIONS:
Drug: Vasopressin Steroids Epinephrine — Vasopressin Steroids Epinephrine: Vasopressin (up to 5 doses of 20 IU) and methylprednisolone (single dose - 40 mg) in addition to epinephrine during cardiopulmonary resuscitation, and stress dose hydrocortisone (300 mg/day for 7 days maximum followed by gradual taper) for postresuscitation shock.
  Other Names: VSE
  Groups: Vasopressin Steroids Epinephrine (VSE)

SUMMARY:
Early stress-dose steroids are of uncertain efficacy in cardiac arrest. The current authors plan to conduct a pertinent mediation analysis using prospectively collected data from 2 prior randomized clinical trials of in-hospital cardiac arrest. These trials reported positive results on the vasopressin-steroids-epinephrine (VSE) combination. The current analysis is aimed at identifying mediators of the benefit associated with VSE, potentially attributable to its stress-dose steroid subcomponent. Tested mediators will include arterial pressure in the early postresuscitation period (primary), and arterial blood lactate in the early postresuscitation period and renal failure free days (secondary).

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE The usefulness of stress-dose hydrocortisone in cardiac arrest is uncertain, especially when its administration starts at 10 hours after the return of spontaneous circulation (ROSC) (1). Such delay, probably exceeds the therapeutic window for the prevention of detrimental episodes of postresuscitation hypotension (2) through a steroid-induced hemodynamic stabilization (3,4).

In the context of NCT02408939, recent post hoc exploratory analyses in postresuscitation shock (n=191) showed an improved early post-ROSC hemodynamic profile in patients treated with the vasopressin-steroids-epinephrine (VSE) combination. Pooled data originated from our prior VSE 1 and VSE 2 randomized clinical trials (RCTs) (3,4) Recordings of "early post-ROSC systolic arterial pressure (SAP) >90" mmHg [i.e. "absence of early postresuscitation hypotension" (2)], and "≥1 recorded/analyzed, day-1 mean arterial pressure (MAP) value of >80mmHg (2)," were significantly more frequent in VSE patients vs. controls. After considering the short vasopressin half-life of 24 min and that the VSE protocol mandates vasopressin use solely during cardiopulmonary resuscitation (CPR) (3,4), we postulate that the more frequent "day-1 MAP>80 mmHg" can be attributed to the MAP-stabilizing effects of early stress-dose steroids (3,4). Under this assumption, a mediation analysis of VSE outcome benefits through day-1 MAP might further address the knowledge gap of steroids' usefulness in cardiac arrest (5).

METHODS Study Design. Intention-to-treat, retrospective analysis of prospectively collected data from two RCTs (3,4). Study participants were hospitalized in intensive or coronary care units (ICUs or CCUs) of three tertiary care centers: Evaggelismos General Hospital and 401 Greek Army Hospital (both in Athens, Greece), and University Hospital of Larissa, Larissa, Greece.

Ethics and Approval. The present analysis of de-identified, previously collected and electronically stored patient data (see also Detailed Descriptions of NCT00729794 and NCT02408939) is not associated with any clinical intervention, and therefore, the investigators have applied for a waiver of informed consent from either the patient or his/her next of kin.

Analysis Endpoints are presented in the dedicated subsection. Patients. The reference study population consists of 368 patients (Evaggelismos Hospital, n=288/368=78.2%) with in-hospital cardiac arrest, who required epinephrine during CPR according to the 2005 Guidelines for Resuscitation (6). During CPR, VSE group patients (n=178) also received vasopressin and methylprednisolone and controls (n=190) the respective saline placebos. At 4 hours after CPR, there were 211 surviving patients (VSE group, n=115), who were evaluated for postresuscitation shock (3,4). One hundred three VSE group patients were then assigned to stress-dose hydrocortisone and 88 controls to saline placebo. Of the 103 VSE group patients, 102 received stress-dose hydrocortisone, whereas 1 did not because of study pharmacist error; of the 88 control group patients, 73 actually received saline placebo, whereas 15 received open-label stress-dose hydrocortisone by protocol violation and according to the orders of their attending physicians (4).

Multivariable Analysis - Effect Modifiers In addition to variables described in the Outcomes subsection, the multivariable analysis will include the following potential effect modifiers: Data Source (VSE2 vs. VSE1 study), Study Center (4), group (VSE vs, control), cardiac arrest cause (cardiac vs. non-cardiac), area of cardiac arrest occurrence (monitored vs. non-monitored), initial cardiac arrest rhythm (shockable vs. non-shockable) atropine use (yes vs. no), prescribed total dose of sodium bicarbonate, cardiac arrest occurrence on holiday vs. working day; Cardiac arrest occurrence at night (23:00-07:00) vs. morning-to-late evening (07:00-23:00), total dose of epinephrine during CPR, and therapeutic hypothermia (use vs. no use).

All analyses will be conducted with SPSS version 22.0 (IBM, Armonk, NY) and the Process Procedure for SPSS, release 2.15. Statistical methodology reference: Hayes AF. Part II, Mediation Analysis. In: Hayes AF, ed. Introduction to Mediation, Moderation, and Conditional Process Analysis. A Regression-based Approach. The Guilford Press, New York. 2013, 3-419. 85-207.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with vasopressor-requiring inhospital cardiac arrest according to guidelines for resuscitation 2005, defined as:

* epinephrine requirement for ventricular fibrillation/tachycardia
* or asystole, or
* pulseless electrical activity

Exclusion Criteria:

* Age < 18 years;
* Terminal illness or do-not resuscitate status;
* Cardiac arrest due to exsanguination;
* Cardiac arrest before hospital admission;
* Pre-arrest treatment with intravenous corticosteroids;
* Previous enrollment in or exclusion from the 2 studies included in the analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with vasopressor-requiring, inhospital cardiac arrest, i.e., with asystole, pulseless electrical activity, or ventricular fibrillation/pulseless ventricular tachycardia not responsive to two attempts at defibrillation. Patients have already participated in 2 prior RCTs (references 3 and 4). Thus, the below-provided Eligibility Criteria are the Criteria already employed by the prior RCTs.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Early postresuscitation systolic arterial pressure (SAP) as mediator of observed intervention benefit. | 20 min after return of spontaneous circulation (ROSC)
  Determination of the possible mediating role of SAP with respect to the observed vasopressin-steroids-epinephrine (VSE) outcome benefit. Multivariable mediation analysis of the following possible relationship: VSE intervention - postresuscitation SAP>90 mmHg at 20 min post-ROSC - Survival with good neurological recovery i.e. Cerebral Performance Category (CPC) score of 1 or 2.This will result in the primary mediation analysis "SAP" model.
Early postresuscitation mean arterial pressure (MAP) as mediator of observed intervention benefit | 24 hours after ROSC
  Determination of the possible mediating role of MAP with respect to the observed VSE outcome benefit. Multivariable mediation analysis of the following possible relationship: VSE intervention - at least 1 day-1 postrandomization MAP value>80 mmHg - Survival with good neurological recovery i.e. CPC score of 1 or 2. This will result in the primary mediation analysis "MAP" model.

SECONDARY OUTCOMES:
Renal failure free days and SAP | Days 1-60 after ROSC
  Addition of renal failure free days to the primary mediation analysis "SAP" model - this will result in a first "multiple mediator" SAP model.
Renal failure free days and MAP | Days 1-60 after ROSC
  Addition of renal failure free days to the primary mediation analysis "MAP" model - this will result in a first "multiple mediator" MAP model.
Arterial blood lactate level > 4.65 mmol/L at 4 hours post-ROSC and SAP | 4 hours post-ROSC
  Addition of arterial blood lactate at 4 hours post-ROSC > 4.65 mmol/L (median value in 191 patients) to the first "multiple mediator" SAP model - this will result in the second "multiple mediator" SAP model.
Arterial blood lactate level > 4.65 mmol/L at 4 hours post-ROSC and MAP | 4 hours post-ROSC
  Addition of arterial blood lactate at 4 hours post-ROSC > 4.65 mmol/L (median value in 191 patients) to the first "multiple mediator" MAP model - this will result in the second "multiple mediator" MAP model.
Arterial blood lactate level > 2.80 mmol/L at 4 hours post-ROSC and SAP | 4 hours post-ROSC
  Addition of arterial blood lactate at 4 hours post-ROSC > 2.80 mmol/L (lower bound of interquartile range in 191 patients) to the first "multiple mediator" SAP model - this will result in the third "multiple mediator" SAP model.
Arterial blood lactate level > 2.80 mmol/L at 4 hours post-ROSC and MAP | 4 hours post-ROSC
  Addition of arterial blood lactate at 4 hours post-ROSC > 2.80 mmol/L (lower bound of interquartile range in 191 patients) to the first "multiple mediator" MAP model - this will result in the third "multiple mediator" MAP model.

CONTACTS AND LOCATIONS:
Overall Officials: Spyros D. Mentzelopoulos, MD, PhD, Principal Investigator — University of Athens; Spyros G. Zakynthinos, MD, PhD, Study Chair — University of Athens
Locations (3):
- Greece (3):
  - Evaggelismos General Hospital, Athens, Attica
  - 401 General Military Hospital of Athens, Athens, Attica
  - Larisa University General Hospital, Larissa, Thessaly

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donnino MW, Andersen LW, Berg KM, Chase M, Sherwin R, Smithline H, Carney E, Ngo L, Patel PV, Liu X, Cutlip D, Zimetbaum P, Cocchi MN; Collaborating Authors from the Beth Israel Deaconess Medical Center's Center for Resuscitation Science Research Group. Corticosteroid therapy in refractory shock following cardiac arrest: a randomized, double-blind, placebo-controlled, trial. Crit Care. 2016 Apr 3;20:82. doi: 10.1186/s13054-016-1257-x. PMID 27038920
- [Background] Trzeciak S, Jones AE, Kilgannon JH, Milcarek B, Hunter K, Shapiro NI, Hollenberg SM, Dellinger P, Parrillo JE. Significance of arterial hypotension after resuscitation from cardiac arrest. Crit Care Med. 2009 Nov;37(11):2895-903; quiz 2904. doi: 10.1097/ccm.0b013e3181b01d8c. PMID 19866506
- [Background] Mentzelopoulos SD, Zakynthinos SG, Tzoufi M, Katsios N, Papastylianou A, Gkisioti S, Stathopoulos A, Kollintza A, Stamataki E, Roussos C. Vasopressin, epinephrine, and corticosteroids for in-hospital cardiac arrest. Arch Intern Med. 2009 Jan 12;169(1):15-24. doi: 10.1001/archinternmed.2008.509. PMID 19139319
- [Background] Mentzelopoulos SD, Malachias S, Chamos C, Konstantopoulos D, Ntaidou T, Papastylianou A, Kolliantzaki I, Theodoridi M, Ischaki H, Makris D, Zakynthinos E, Zintzaras E, Sourlas S, Aloizos S, Zakynthinos SG. Vasopressin, steroids, and epinephrine and neurologically favorable survival after in-hospital cardiac arrest: a randomized clinical trial. JAMA. 2013 Jul 17;310(3):270-9. doi: 10.1001/jama.2013.7832. PMID 23860985
- [Background] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995
- [Background] Nolan JP, Deakin CD, Soar J, Bottiger BW, Smith G; European Resuscitation Council. European Resuscitation Council guidelines for resuscitation 2005. Section 4. Adult advanced life support. Resuscitation. 2005 Dec;67 Suppl 1:S39-86. doi: 10.1016/j.resuscitation.2005.10.009. No abstract available. PMID 16321716